CLINICAL TRIAL: NCT04296825
Title: Effect of Camel Milk Containing Bifidobacterium Animalis A6 on Chinese People With Type 2 Diabetes Mellitus
Brief Title: Effect of Camel Milk With Probiotic on Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: China Agricultural University (Other)
Collaborators: Beijing Chinese Medicine Hospital-Pinggu Hospital (Unknown)
Responsible Party: Principal Investigator, Fazheng Ren, Professor, China Agricultural University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FDLT2DM-01
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2018-06

CONDITIONS: Type 2 Diabetes
Keywords: Camel Milk; Probiotics; Gut Microbiome
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- P (Placebo Comparator): Patients received cow milk for 4 consecutive weeks (two times per day, 10 gram each time).
  Interventions: Dietary Supplement: Cow milk
- CA (Active Comparator): Patients received camel milk with Bifidobacterium animalis A6 at a dose of 2×1010 viable cells for 4 consecutive weeks (two times per day, 10 gram each time).
  Interventions: Dietary Supplement: Camel milk containing Bifidobacterium animalis A6
- C (Experimental): Patients received camel milk for 4 consecutive weeks (two times per day, 10 gram each time).
  Interventions: Dietary Supplement: Camel milk
- A (Experimental): Patients received Bifidobacterium animalis A6 at a dose of 2×1010 viable cells for 4 consecutive weeks (two times per day, 10 gram each time).
  Interventions: Dietary Supplement: Bifidobacterium animalis A6

INTERVENTIONS:
Dietary Supplement: Camel milk containing Bifidobacterium animalis A6 — Take the interventions about 30 minutes after meals in the morning and evening for 4 consecutive weeks.
  Arms: CA
Dietary Supplement: Camel milk — Take the interventions about 30 minutes after meals in the morning and evening for 4 consecutive weeks.
  Arms: C
Dietary Supplement: Bifidobacterium animalis A6 — Take the interventions about 30 minutes after meals in the morning and evening for 4 consecutive weeks.
  Arms: A
Dietary Supplement: Cow milk — Take the interventions about 30 minutes after meals in the morning and evening for 4 consecutive weeks.
  Arms: P

SUMMARY:
The purpose of this study is to investigate the effects of dietary supplement with Camel Milk containing Bifidobacterium animalis A6 on the plasma glucose and other related cytokines in patients with type 2 diabetes mellitus. 45 patients with type 2 diabetes mellitus were recruited, and a Double Blind Randomized Parallel Controlled Trial was performed. The fasting glycaemia, 2 hour postprandial glycaemia, insulin, uric acid and serum lipid (total cholesterol, total triglyceride, high-density lipoprotein cholesterol and low-density lipoprotein cholesterol ) were measured as Primary Outcome. The Fecal microbiome, fecal metabolites, gut hormones (amylin, ghrelin, glucagon-like peptide 1, pancreatic polypeptide), inflammation cytokines (TNF-α, IL-6, MCP-1), myokines (FGF-21, irisin, osteocrin/musclin, osteonectin) and adipokines (adiponectin, resistin, lipocalin-2, adipsin) and body composition analysis were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35~68 years old
* Patients who diagnosed as type 2 diabetes
* Agree to take the products to be studied during the study period, and no longer take other fermented dairy products (live lactic acid bacteria drinks, cheese, yogurt, probiotic products, etc.) and antibiotic
* Agree to sign the informed consent form

Exclusion Criteria:

* Taking antibiotics or antifungal drugs within 7 days before the study
* Have serious allergic reaction to skim milk powder or milk
* Researcher are not sure whether the subjects are willing or able to complete the study
* Subject had other serious diseases

Ages: 35 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-06-09 (Actual); Study Completion 2018-07-09 (Actual)

PRIMARY OUTCOMES:
Changes in fasting blood glucose and 2 hour postprandial blood glucose in millimole per liter and insulin in μU/mL | 4 weeks
  follow up the patients at week 0, 4
Changes in lipid profiles (total cholesterol, total triglyceride, high-density lipoprotein cholesterol and low-density lipoprotein cholesterol in millimole per liter) | 4 weeks
  follow up the patients at week 0, 4

SECONDARY OUTCOMES:
Changes in inflammation cytokines ( TNF-α, IL-6 and MCP-1 in petagram per milliliter) | 4 weeks
  follow up the patients at week 0, 4
Changes in fecal microbiome | 4 weeks
  follow up the patients at week 0, 4
Fecal metabolites were identified by GC-MS after extracted with methanol, then oximated with methoxyamine hydrochloride and trimethylsilylated with BSTFA. The concentration was calculated as the area of the peak and normalized to the internal standard. | 4 weeks
  follow up the patients at week 0, 4
Changes in body composition (bodyweight in kilograms, height in meters and visceral fat content in square centimeters and body fat in % were measured using the bioelectrical impedance method (BAS-H, SEEHIGHER, Beijing China). ) | 4 weeks
  follow up the patients at week 0, 4
Changes in myokines (FGF21, irisin, osteocrin, and osteonectin in petagram per milliliter) and adipokines (adiponectin and adipsin in microgram per milliliter and resistin and lipocalin-2 in petagram per milliliter) | 4 weeks
  follow up the patients at week 0, 4
Changes in gut hormones (amylin, ghrelin, GLP-1, PP and PYY in petagram per milliliter) | 4 weeks
  follow up the patients at week 0, 4

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chinese Medicine Hospital Pinggu Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auer HE, Doty P. The synthesis, structure, and optical properties of some copolypeptides containing nonpolar amino acid residues. Biochemistry. 1966 May;5(5):1708-15. doi: 10.1021/bi00869a037. No abstract available. PMID 5961288
- [Result] Agrawal RP, Budania S, Sharma P, Gupta R, Kochar DK, Panwar RB, Sahani MS. Zero prevalence of diabetes in camel milk consuming Raica community of north-west Rajasthan, India. Diabetes Res Clin Pract. 2007 May;76(2):290-6. doi: 10.1016/j.diabres.2006.09.036. Epub 2006 Nov 13. PMID 17098321
- [Result] Saigusa M, Mizuno A, Morimoto K, Nakamura K. [Acute postoperative renal failure due to extracorporeal circulation--with reference to the evaluation of fatal cases]. Kyobu Geka. 1967 Sep;20(9):594-9. No abstract available. Japanese. PMID 5626114
- [Result] Casini F, Sbarigia V, Schiavone C. [Identification of Cannabis indica in the residues of incomplete combustion of the drug]. Boll Chim Farm. 1969 May;108(5):330-6. No abstract available. Italian. PMID 5806827
- [Result] Baumgarten A, Melrose GJ, Vagg WJ. Continuous recording of dermal exudative reactions. Dermatologica. 1970;140(4):219-24. doi: 10.1159/000252557. No abstract available. PMID 5425915
- [Result] Burdon JF. [Medicine in Great Britain]. Concours Med. 1965 Oct 9;87(41):5799-803. No abstract available. French. PMID 5857053
- [Result] Lavin MF, Seymour GJ. Reduced levels of fibronectin in ataxia-telangiectasia lymphoblastoid cells. Int J Cancer. 1984 Mar 15;33(3):359-63. doi: 10.1002/ijc.2910330313. PMID 6365801